CLINICAL TRIAL: NCT03529396
Title: Safety and Efficacy of Different Regimens of Primaquine on Vivax Malaria Treatment in Glucose 6-phosphate Dehydrogenase Deficient Patients
Brief Title: Safety and Efficacy of Different Regimens of Primaquine on Vivax Malaria Treatment in G6PD Deficient Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Oswaldo Cruz Foundation (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Wuelton Marcelo Monteiro, PhD, Director of Research, Fundação de Medicina Tropical Dr. Heitor Vieira Dourado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 70177317.1.0000.0005
Record Dates: First submitted 2018-04-25; First posted 2018-05-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Vivax Malaria; G6PD Deficiency
Keywords: G6PD deficiency; Acute hemolytic anemia; Vivax malaria; Primaquine; Weekly primaquine; Chloroquine; Weekly chloroquine; Brazilian Amazon; Oxidative stress
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1a: Chloroquine + 5th-day Primaquine (Experimental): [ARM HALTED PREMATURELY DUE TO SAFETY CONCERNS]
  Interventions: Drug: Chloroquine; Drug: Primaquine
- 1b: Chloroquine + 8-week Primaquine (Experimental): 26 G6PD deficient patients. Directly observed therapy.
  Interventions: Drug: Chloroquine; Drug: Primaquine
- 1c: Chloroquine + 12-week Chloroquine (Active Comparator): 26 G6PD deficient patients. Control group in terms of safety. Directly observed therapy.
  Interventions: Drug: Chloroquine
- 2: Standard chloroquine + primaquine (Active Comparator): 52 G6PD normal patients. Control group in terms of efficacy. Directly observed therapy.
  Interventions: Drug: Chloroquine; Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine — Standard chloroquine (three days)
Drug: Primaquine — Daily Primaquine (0.5 mg of base/kg/day for seven days) starting only at the fifth day post chloroquine initiation.
  Arms: 1a: Chloroquine + 5th-day Primaquine
Drug: Primaquine — Weekly primaquine (0.75 mg of base/kg/week for eight weeks) starting with first dose of chloroquine.
  Arms: 1b: Chloroquine + 8-week Primaquine
Drug: Chloroquine — Weekly, once a week chloroquine (5 mg of base/kg/week for twelve weeks)
  Arms: 1c: Chloroquine + 12-week Chloroquine
Drug: Primaquine — Standard primaquine (0.5mg of base/kg/day for seven days) concomitant with chloroquine.
  Arms: 2: Standard chloroquine + primaquine

SUMMARY:
A clinical study to assess the safety and efficacy of alternative regimens of primaquine for radical cure of vivax malaria in glucose 6-phosphate dehydrogenase (G6PD) deficient. G6PD deficient patients with P. vivax monoinfection will be treated with either weekly or delayed one-week course of primaquine, and the currently recommended by national guideline, 12-week chloroquine regimen to compare treatment safety among groups. All groups will be actively monitored for hemolysis during treatment and will have six-month follow-up period to assess treatment efficacy.

DETAILED DESCRIPTION:
This is an open-label, randomized, phase II, clinical trial of safety and efficacy. Patients will be screened for eligibility and treated at the Fundação de Medicina Tropical Dr Heitor Vieira Dourado in Manaus and the Centro de Pesquisa em Medicina Tropical (Cepem) in Porto Velho, Brazil. A total of 104 vivax malaria patients will be recruited into the study, 52 G6PD deficient (Arm 1) and 52 G6PD normal (Arm 2). Patients with spectrophotometrically-confirmed G6PD deficiency (10-60% of adjusted mean male activity) will be divided into three subgroups of 10 patient each. All arms will receive standard 3-day chloroquine course. Additionally, Arm 1a will receive a delayed course of primaquine for 7 days, starting only at the fifth-day post-chloroquine initiation [ARM HALTED DUE TO SAFETY CONCERNS]. Arm 1b will receive weekly primaquine, once a week, for 8 weeks. Arm 1c will receive prophylactic 12-week course of chloroquine, as recommended by national guidelines for such patients (control group in terms of safety). Arm 2, the control group of efficacy, will receive standard regimen, comprised of 3-day chloroquine plus concomitant 7-day primaquine. All patients will receive directly observed therapy (DOT) and will be closely monitored for clinical parameters and laboratory markers of hemolysis including hemoglobin, methemoglobin, lactate dehydrogenase, haptoglobin, reticulocytes, indirect bilirubin, aspartate aminotransferase, and urinalysis. All groups will be followed for 6 months after treatment to assess relapse rate. Primary endpoint is the tolerability of the regimens defined by hemoglobin fall. Secondary endpoints include treatment failure (relapse during follow-up), frequency of adverse effects, and rate of hemoglobin fall during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated vivax malaria monoinfection
* G6PD deficiency ranging from 10%-60% of adjusted mean male activity
* Baseline hemoglobin >9 g/dL
* Willing to comply with study requirements

Exclusion Criteria:

* Pregnancy or breastfeeding
* Comorbidities (hepatopathy and/or nephropathy)
* Use of antimalarials in the previous two weeks or current use of potentially hemolytic drugs
* Any condition which would place the subject at undue risk of hemolysis or interfere with the results of the study, as judged by investigator.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Absolute or relative change in hemoglobin < 3g/dL or 30% from baseline | From date of randomization until the date of last dose, assessed up to 12 weeks.
  Hemoglobin reduction from baseline after exposure to primaquine for P. vivax treatment

SECONDARY OUTCOMES:
Regimen efficacy | 6 months post treatment
  Relapse rate over follow-up period after treatment
Adverse effects | From date of randomization until the date of first documented event, assessed up to 12 weeks.
  Presence of adverse reactions as a result of intervention, measured by clinical and laboratory tests
Change in hemoglobin values over treatment | through study completion: before intervention and up to 12 weeks during intervention.
  Absolute variation of hemoglobin levels before and during intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus VG Lacerda, MD, PhD, Principal Investigator — Fiocruz/ILMD and Fundacao de Medicina Tropical Dr Heitor Vieira Dourado
Locations (2):
- Brazil (2):
  - Fundação de Medicina Tropical Doutor Heitor Vieira Dourado, Manaus, Amazonas
  - Centro de Pesquisa em Medicina Tropical (Cepem), Porto Velho, Rondônia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barbosa L, Brito-Sousa J, Nascimento C, Pacheco A, Alexandre M, Alencar A, Melo M, Omena A, Souza I, Silva E, Queiroz M, Siqueira V, Rabelo C, Baia-da-Silva D, Silva D, Rocha Y, Barbosa A, Castro R, Almeida A, Brito M, Lopes A, Balieiro A, Costa M, Amaral T, Valle C, Vieira A, Gonzaga J, Pereira D, Alecrim M, Monteiro W, Lacerda M, Melo G. Safety and Efficacy of 3 Alternative Regimens Against Relapsing Plasmodium vivax Malaria in Glucose 6-Phosphate Dehydrogenase-Deficient Patients in the Brazilian Amazon (ALTPRIM). Clin Infect Dis. 2025 Dec 24;81(5):e294-e301. doi: 10.1093/cid/ciaf007. PMID 39785834